CLINICAL TRIAL: NCT03227913
Title: Evaluate the Link Between the Characteristics of Oral Physiology and the Formation of the Food Bolus During the Consumption of Cheese Products in Elderly People
Brief Title: Evaluate the Link Between the Characteristics of Oral Physiology and the Formation of the Food Bolus During the Consumption of Dairy Products in Elderly People
Acronym: AlimaSSenSLait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VVW Alimassens lait ANR 2014
Record Dates: First submitted 2017-06-26; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Old Person

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good chewing ability (Active Comparator)
  Interventions: Other: Two samples of saliva; Other: Chewing behaviour; Other: Study of the food bolus
- Impaired chewing ability (Experimental)
  Interventions: Other: Two samples of saliva; Other: Chewing behaviour; Other: Study of the food bolus

INTERVENTIONS:
Other: Two samples of saliva — 1. Without stimulation: the first will be used to measure the flow of naturally secreted saliva
  2. With stimulation: the second will will be used to measure the flow and viscosity of the saliva secreted after stimulation
Other: Chewing behaviour — Measure the time taken by subjects to chew the food and the number of bites they use before swallowing
Other: Study of the food bolus — * Analysis by a compression and viscosity test
  * Evaluation of the quantity of saliva incorporated by drying

SUMMARY:
The aim of this study is to understand how dairy products enriched in minerals and proteins are broken down in the mouth. More specifically, investigators wish to evaluate the link between oral physiology (salivation and mastication) and formation of the food bolus during the consumption of enriched cheese, that is to say the way in which the food is broken down to be swallowed.

The study will take place at the INRA in Dijon during 2 one-hour sessions spread over 4 months. These two sessions will allow investigators to characterise the chewing behaviour of the subjects and their salivation, and the structure of the food bolus formed when eating the four products of the project.

For each of the four foods in each session:

* Two samples of saliva will be taken
* A video will be made of subjects eating one of the study products
* Subjects will chew the study foods and spit them out.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written consent
* Age ≥ 65 years old
* Persons living at home
* Persons who can travel independently

Exclusion Criteria:

* Adults under guardianship
* Persons without health insurance cover
* Persons in hospital
* Persons in institutions
* Persons whose Mini-Mental State Examination (MMSE) is < 24
* Persons requiring enteral or parenteral nutrition
* Persons who in the previous 12 months received € 4500 for taking part in clinical trials, including the present study
* Persons in a period of exclusion of a previous study
* Food allergies (dairy products in particular)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Duration of chewing | Change from baseline at 4 months
Frequency of chewing | Change from baseline at 4 months
Rheology test | Change from baseline at 4 months
calculation of insanity rate | Change from baseline at 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France